CLINICAL TRIAL: NCT01511393
Title: Medullary Thyroid Carcinoma Surveillance Study: A Case-Series Registry
Brief Title: An Active Surveillance Program for Cases of Medullary Thyroid Carcinoma (MTC)
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Collaborators: AstraZeneca (Industry); Eli Lilly and Company (Industry); United BioSource, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3965; U1111-1125-4362 (Other: WHO)
Record Dates: First submitted 2011-11-30; First posted 2012-01-18 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Medullary Thyroid Carcinoma; Weight Management
Keywords: GLP1; Glucagon like peptide; liraglutide; exenatide extended release; dulaglutide; semaglutide; semaglutide tablets
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Questionnaire: None. Non-interventional study.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — None. Non-interventional study.

SUMMARY:
This study is conducted in the United States of America (USA). The aim of the study is to monitor the number of annual new adult cases of medullary thyroid carcinoma (MTC) and to establish a registry for these new cases in order to identify any possible increase related to the introduction of liraglutide, exenatide once-weekly, and other GLP-1 receptor agonists into the US market.

DETAILED DESCRIPTION:
This active surveillance program will monitor for any signal indicating a possible association between treatment with long-acting GLP-1 RAs and the development of MTC in the United States population. Given the very low incidence of MTC in the general population, the expected rate of exposure to long-acting GLP-1 RAs, the anticipated long latency of the potential outcome under study and the limited data on underlying risk factors for development of MTC other than RET proto-oncogene mutations, an active surveillance program is the most efficient means of identifying a possible association between MTC and products in the long-acting GLP-1 RAs class. Given the uncertainty of the association of MTC in humans treated with these drugs, a study duration of at least fifteen years from the time of market introduction of the first long-acting GLP-1 RA was thought to provide evidence of an association, if one exists. If such an association is identified, a case-control study will be initiated to quantify the association.

The MTC registry is a Food and Drug Administration (FDA) post-marketing requirement for long-acting GLP-1 RA products. Because of the rarity of MTC and in order to minimize inconvenience to patients, physicians, and state cancer registries, FDA encouraged sponsors of long-acting GLP-1 RAs to work collaboratively to conduct this registry. Consequently, the MTC Registry Consortium has been formed for this purpose.

The MTC Registry Consortium refers to the Sponsors with approved long-acting GLP-1 RAs who have a contractual agreement to participate in the MTC Registry.

This active surveillance program for cases of MTC will be conducted with assistance from the North American Association of Central Cancer Registries (NAACCR). NAACCR is a collaborative umbrella organization for cancer registries, government agencies, professional organizations, and private groups in North America interested in improving the quality and use of cancer registry data. All of the central cancer registries in the U.S. and Canada are members of NAACCR, including those that participate in SEER.

ELIGIBILITY:
Inclusion Criteria:

* A record of medullary thyroid carcinoma (MTC) identified from state/regional population-based cancer registries
* At least 18 years or older.

There are no other inclusion or exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with medullary thyroid carcinoma invited by either written invitation from the participating cancer registry or the diagnosing physician to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 6750 (Estimated)
Dates: Start 2012-01; Primary Completion 2039-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Annual incidence of MTC in the US to identify any possible increase related to the introduction of liraglutide, exenatide once-weekly, and other GLP-1 receptor agonists into the US market. | Up to 15 years

SECONDARY OUTCOMES:
Family history of cancer (including history of MEN2A or MEN 2B, history of FMTC, history of RET proto-oncogene mutations), Patient demographic characteristics, Patient prior history of thyroid diseases | Up to 15 years
Dose and Duration of use of all previous diabetes medication exposures (including long acting and short acting GLP-1 receptor agonists, DPP4 inhibitors, and insulin) | Up to 15 years
Dose and Duration of use of all previous weight management drugs (including long acting GLP-1 receptor agonists). | Up to 15 years
Lifestyle factors such as smoking and alcohol use | Up to 15 years
Environmental exposures (occupational history, radioiodine exposure, nuclear fallout) | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Annette Stemhagen, DrPH, FISPE, Study Director — United BioSource, LLC
Locations (1):
- United BioSource, LLC, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Currently this is undecided for this 15 year registry. The Data Monitoring Committee is a group of external interdisciplinary consultants who oversee the registry data to review if there are any signals or safety concerns with patients who have taken any of the long-acting GLP-1 RAs and were diagnosed with medullary thyroid carcinoma.

REFERENCES:
- [Derived] Major-Pedersen A, McCullen MK, Sabol ME, Adetunji O, Massaro J, Neugut AI, Sosa JA, Hollenberg AN. A joint industry-sponsored data monitoring committee model for observational, retrospective drug safety studies in the real-world setting. Pharmacoepidemiol Drug Saf. 2021 Jan;30(1):9-16. doi: 10.1002/pds.5172. Epub 2020 Nov 24. PMID 33179845
- See also: AstraZeneca Pharmaceuticals LP — http://astrazenecagrouptrials.pharmacm.com/